CLINICAL TRIAL: NCT02280018
Title: A Double Blind, Placebo-Controlled, Randomized Study to Investigate the Safety, Tolerability, and Pharmacokinetics of a Single Intravenous Dose of JNJ-49122944 in Healthy Male Subjects
Brief Title: A Safety, Tolerability and Pharmacokinetics Study of a Single Intravenous Dose of JNJ-49122944 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR105925; 49122944EDI1001 (Other: Janssen Research & Development, LLC); 2014-002354-39 (EudraCT Number)
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: Healthy; JNJ-49122944; Placebo

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- JNJ-49122944, 5 milligram (mg) (Experimental): Single dose of 5 mg JNJ-49122944, administered as a 22.2 milliliter (mL) intravenous (IV) infusion over 45 minutes in the morning following an overnight fast.
  Interventions: Drug: JNJ-49122944, 5 milligram (mg)
- Placebo (Placebo Comparator): Placebo matched to JNJ-49122944, administered as a 22.2 mL IV infusion over 45 minutes in the morning following an overnight fast.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-49122944, 5 milligram (mg) — Participants will receive single dose of 5 mg JNJ-49122944, administered as a 22.2 mL IV infusion over 45 minutes on Day 1.
  Arms: JNJ-49122944, 5 milligram (mg)
Drug: Placebo — Participants will receive placebo matched to JNJ-49122944, administered as a 22.2 mL IV infusion over 45 minutes on Day 1.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics (the study of the way a drug enters and leaves the blood and tissues over time) of JNJ-49122944 in healthy male participants after a single intravenous ([IV] within a vein) dose administration.

DETAILED DESCRIPTION:
This is a double-blind (neither the researchers nor the participants know what treatment the participant is receiving), randomized (study drug assigned by chance), placebo-controlled (an inactive substance; a pretend treatment [with no drug in it] that is compared in a clinical trial with a drug to test if the drug has a real effect), and single-center study. The study will consist of Screening Period (2 to 21 days prior to participants' dose administration), Double-blind Treatment Period (single dose of JNJ-49122944 or placebo on Day 1), and Safety Follow-up Period (4 to 7 days after discharge). The total duration of participation for each participant, including screening, will be up to approximately 4 weeks. Blood samples will be collected for assessment of pharmacokinetic parameters. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male participant, aged 18 to 55 inclusive
* Participant must have a body Mass Index (BMI) between 18 and 30 kilogram per square meter (kg/m^2), inclusive, and body weight not less than 50 kg
* Participant must be deemed healthy on the basis of physical examination, medical history, laboratory tests, vital signs, and 12-lead electrocardiogram within protocol-defined parameters performed at screening and Day -1
* Participant agrees to protocol-defined use of effective contraception
* Participant should be non-nicotine user for 6 months prior to screening

Exclusion Criteria:

* Participants with current or history of clinically significant medical illness
* Participants with history of drug or alcohol abuse within 5 years
* Routine consumption of greater than 450 milligram (mg) of caffeine per day by the participant
* Participants with recent vaccination or acute illness
* Blood donation or major blood loss within 3 months prior to study drug administration by the participant

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) | Throughout the duration of study (up to 4 weeks)
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Maximum Plasma Concentration (Cmax) of JNJ-49122944 | Pre-dose, 0.25, 0.50, 0.75, 1, 1.25, 1.75, 2.75, 4.75, 6.75, 12.75 hour post- dose on Day 1, 24.75 hour post-dose on Day 2, 48.75 hour post-dose on Day 3
  The Cmax is the maximum observed plasma concentration during dosing interval.
Area Under the Plasma Concentration Time Curve From Time 0 to Last Quantifiable Time (AUClast) of JNJ-49122944 | Pre-dose, 0.25, 0.50, 0.75, 1, 1.25, 1.75, 2.75, 4.75, 6.75, 12.75 hour post- dose on Day 1, 24.75 hour post-dose on Day 2, 48.75 hour post-dose on Day 3
  The AUC(last) is the area under the plasma concentration time curve from time 0 to the time corresponding to the last quantifiable plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of JNJ-49122944 | Pre-dose, 0.25, 0.50, 0.75, 1, 1.25, 1.75, 2.75, 4.75, 6.75, 12.75 hour post- dose on Day 1, 24.75 hour post-dose on Day 2, 48.75 hour post-dose on Day 3
  The AUC(0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Percentage of Area Under the Plasma Concentration-time Curve Obtained by Extrapolation (%AUC [infinity,ex]) of JNJ-49122944 | Pre-dose, 0.25, 0.50, 0.75, 1, 1.25, 1.75, 2.75, 4.75, 6.75, 12.75 hour post- dose on Day 1, 24.75 hour post-dose on Day 2, 48.75 hour post-dose on Day 3
  Percentage of area under the plasma concentration-time curve obtained by extrapolation (%AUC[inf,ex]) is calculated by dividing the difference of AUC(0-infinity) and AUC(0-last) by AUC(0-infinity) and then multiplying by 100 (AUC[0-infinity] - AUC[0-last])*100/AUC[0-infinity].
Elimination Half-life (t1/2) of JNJ-49122944 | Pre-dose, 0.25, 0.50, 0.75, 1, 1.25, 1.75, 2.75, 4.75, 6.75, 12.75 hour post- dose on Day 1, 24.75 hour post-dose on Day 2, 48.75 hour post-dose on Day 3
  Elimination half-life (t [1/2]) is associated with the terminal slope (lambda [z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Rate Constant (Lambda[z]) of JNJ-49122944 | Pre-dose, 0.25, 0.50, 0.75, 1, 1.25, 1.75, 2.75, 4.75, 6.75, 12.75 hour post- dose on Day 1, 24.75 hour post-dose on Day 2, 48.75 hour post-dose on Day 3
  Lambda(z) is first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Apparent Clearance (CL) of JNJ-49122944 | Pre-dose, 0.25, 0.50, 0.75, 1, 1.25, 1.75, 2.75, 4.75, 6.75, 12.75 hour post- dose on Day 1, 24.75 hour post-dose on Day 2, 48.75 hour post-dose on Day 3
  Apparent clearance of JNJ-49122944 is calculated as Dose/AUC(infinity). The AUC (infinity) is the area under the plasma concentration-time curve from time zero to infinite time.
Apparent Volume of Distribution (Vz) of JNJ-49122944 | Pre-dose, 0.25, 0.50, 0.75, 1, 1.25, 1.75, 2.75, 4.75, 6.75, 12.75 hour post- dose on Day 1, 24.75 hour post-dose on Day 2, 48.75 hour post-dose on Day 3
  Apparent volume of distribution after intravenous administration is calculated as Dose divided by Lambda(z) multiplied by AUC(0-inifinity).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium